CLINICAL TRIAL: NCT03827863
Title: The Prospective Observational Study of ARDS Related Acute CorPulmonale and the Randomized Controlled Study of ARDS Aimed Circulation Protection China (ACPC)
Brief Title: Acute CorPulmonale and ARDS Circulation Protection China Study China (ACPC)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HS-1615
Record Dates: First submitted 2019-01-29; First posted 2019-02-04 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: ARDS (Acute Respiratory Distress Syndrome); Acute Cor Pulmonale
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood specimen, morning blood samples were collected at the baseline assessment and will be collected at the follow-ups. After simple processing, the supernatant was separated after centrifugation and frozen at -80°C at each participating centre, and then transported to the central laboratory by cold chain every 3 months for future use.
  With these specimens, we intend to explore for novel biomarkers that reflect ARDS progression and develop predictive models to identify a subgroup population among ARDS with ACP who are at high risk. Examples of biomarkers to explore include glycocalyx shedding, vascular endothelium, and inflammatory factors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ARDS WITH ACP: 1. Diagnostic criteria for ARDS ARDS defined as within 1 week of a known clinical insult or new or worsening respiratory symptoms. ARDS was classified as mild (200 mmHg < PaO2/FIO2≤300 mmHg), moderate (100 mmHg < PaO2/FIO2≤200 mmHg) and severe (PaO2/FIO2≤100 mmHg) according to the value of PaO2/FiO2 ratio. Importantly, the PaO2/FiO2 ratio value is considered only with a CPAP or PEEP value of at least 5 cmH2O.
  2. Ultrasound diagnostic criteria for ACP The specific diagnostic parameters are as follows: TR>2.8m/s; RVEDA/LVEDA>0.6 or Right ventricle/left ventricle basal diameter ratio>1.0 or systolic D sign; IVC >2cm with decreased inspiratory collapse; Pulmonary Regurgitation Velocity >2.2m/s.
  Interventions: Device: TTE
- ARDS WITHOUT ACP: Diagnosis as ARDS but no ultrasound evidence of ACP.
  Interventions: Device: TTE

INTERVENTIONS:
Device: TTE — TTE to detect the heart function

SUMMARY:
The investigators established a national cohort of Chinese ARDS with Acute CorPulmonale to enable prospective observational studies. The goals are the following.

First, morbidity and mortality rate of ARDS with ACP in the ICU across Chinese mainland.

Second, forming the diagnostic ultrasound strategy of ARDS-ACP, namely TRIP procedures. And predictive value of diagnostic strategy for ACP or prognosis of ACP were calculated.

Third, comparison of ventilator parameters for ACP and non-ACP or survivor and non-survisors, which reaveald that of inappropriate mechanical ventilation on circulation and prognosis. Screening for risk factors of ARDS with ACP.

DETAILED DESCRIPTION:
Acute respiratory distress syndrome (ARDS) is an acute and critical illness characterized by progressive dyspnea and refractory hypoxemia caused by intrapulmonary or extrapulmonary factors. The mortality rate of ARDS is extremely high. ACP caused by pulmonary circulatory disorder is its main clinical feature, which is related to the severity of lung injury in ARDS patients. It has been recognized that the ACP is an independent risk factor for the prognosis of patients with ARDS. Positive pressure mechanical ventilation is an important ARDS treatment strategy for ARDS. Especially the lung protective ventilation strategy with "small tidal volume and increased PEEP" as the core content, which achieved a milestone of lower the mortality of ARDS. However, improper use of positive pressure mechanical ventilation can increase right ventricular load and increase mortality in ARDS patients. Therefore, understanding the effect of positive pressure mechanical ventilation on right heart function in patients with ARDS is important for prevention and treatment for the ACP of ARDS and reduction of ARDS mortality.

The alveolar edema, alveolar collapse, and hypoxic pulmonary vasoconstriction loss caused by increased pulmonary vascular permeability and release of inflammatory mediators resulted in loss of ventilation/blood flow, severe hypoxemia, pulmonary vasospasm, pulmonary microthrombus formation, which increased pulmonary arterial pressure and even APC. Positive pressure mechanical ventilation maintains alveolar ventilation through positive airway pressure, prevents premature alveolar collapse by positive end expiratory pressure (PEEP), changes intrathoracic pressure and lung volume, and affects the right ventricle load. Different studies have found that the incidence of ACP in patients with ARDS is from 22% to 60%. Jardin, et al found that patients with ARDS had a significant increase in ACP and mortality when the airway pressure was greater than 26 cmH2O, which revealed that the difference in positive pressure mechanical ventilation settings has a significant difference in the right heart function of ARDS patients. Mekontso, et al propose a simple clinical risk score for early identification of ACP included pneumonia as cause of ARDS, driving pressure ≥18cmH2O, PaO2/FiO2 ratio<150 mmHg, and PaCO2≥48mmHg. However, for the morbidity and mortality of ACP in ARDS, the related risk factors and criteria are different due to the influence of the different etiology of ARDS and the different study time. For these reasons, the investigators established a national cohort of Chinese ARDS with Acute CorPulmonale to enable prospective observational studies.

ELIGIBILITY:
Inclusion Criteria:

* 18≤ aged ≤85 years old
* received a diagnosis of ARDS with Acute CorPulmonal
* provided signed informed consent

Exclusion Criteria:

* are diagnosed as cardiogenic pulmonary edema
* are diagnosed as Idiopathic pulmonary fibrosis acute exacerbation
* are participating in other interventional clinical trials
* refused to continue to participate in the study or refused further treatment
* unable to complete the study procedure even if assisted and otherwise unable to comply with the study protocol

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the critically patients admitted to ICU
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2020-01-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
28 days SURVIVAL | 28 days after ICU admission
length of stay of ICU | 1 years
mechanical ventilation time | 1 years

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided
When the study begin.

REFERENCES:
- [Derived] Su LX, Shang XL, Zhu R, He W, Pan P, Zhang HM, Zhang LN, Liu DW, Yu RG, Wang XT; Chinese Critical Ultrasound Study Group (CCUSG). A cross-sectional study of acute cor pulmonale in acute respiratory distress syndrome patients in China. Chin Med J (Engl). 2019 Dec 5;132(23):2842-2847. doi: 10.1097/CM9.0000000000000531. PMID 31856056